CLINICAL TRIAL: NCT04780100
Title: Distinguishing Acetabulum Cup Retroversion From Anteversion on Anteroposterior Radiographs After Total Hip Arthroplasty
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Taipei Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: N202005040
Record Dates: First submitted 2021-02-22; First posted 2021-03-03 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2020-07

CONDITIONS: Orthopedics

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this study, investigators will demonstrate and prove a ellipse method (Liaw's version) for measurement and detection of acetabulum cup retroversion.

DETAILED DESCRIPTION:
Total hip arthroplasty (THA) is considered to be the best and most reliable treatment of end-stage hip disorders with satisfactory long-term clinical outcomes. However,the incidence of postoperative dislocation ranges from 0.3% to 3% in primary THA. The most important risk factor is malpositioning of implant components. Generally, excessive anteversion and retroversion increase risk of anterior and posterior hip dislocation respectively. Several radiological methods have been proposed to measure anteversion of the acetabular cup on plain radiographs, but most of these methods cannot accurately distinguish cup retroversion from anteversion. In this study, investigators will demonstrate and prove a ellipse method (Liaw's version) for measurement and detection of acetabulum cup retroversion.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergone total hip arthroplasty
* Patients undergone total hip arthroplasty with more than two postoperative anteroposterior radiographs of pelvis
* Patients undergone total hip arthroplasty with postoperative pelvic CT

Exclusion Criteria:

* Patients with congenital pelvis abnormality or pelvic fracture history
* Patients with postoperative periprosthetic fracture(s)
* Patients with postoperative infection or implants loosening
* Patients undergone total hip arthroplasty without more than two postoperative anteroposterior radiographs of pelvis
* Patients undergone total hip arthroplasty without postoperative pelvic CT

Ages: 30 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients from Shuang Ho Hospital
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2021-03 (Estimated); Primary Completion 2021-05 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
A computerized ellipse method (Liaw's version) for measurement and detection of acetabulum cup retroversion. | 10 days
  Total hip arthroplasty (THA) is considered to be the best and most reliable treatment of end-stage hip disorders with satisfactory long-term clinical outcomes. However,the incidence of postoperative dislocation ranges from 0.3% to 3% in primary THA. The most important risk factor is malpositioning of implant components. Generally, excessive anteversion and retroversion increase risk of anterior and posterior hip dislocation respectively. Several radiological methods have been proposed to measure anteversion of the acetabular cup on plain radiographs, but most of these methods cannot accurately distinguish cup retroversion from anteversion. In this article, we will demonstrate and prove a computerized ellipse method (Liaw's version) for measurement and detection of acetabulum cup retroversion.

CONTACTS AND LOCATIONS:
Overall Officials: Chen-Kun Liaw, Study Chair — Taipei Medical University

IPD SHARING:
Plan to Share IPD: Undecided